CLINICAL TRIAL: NCT06658522
Title: RECOMPENSE: Right vEntricular COMPENsation With SotatercEpt: a Prospective Single Arm Open Label Phase 4 Study to Evaluate the Effects of Sotatercept on Right Ventricular Function in Pulmonary Arterial Hypertension
Brief Title: Right Ventricular Compensation With Sotatercept: A Prospective Single Arm Open Label Phase 4 Study to Evaluate the Effects of Sotatercept on Right Ventricular Function in Pulmonary Arterial Hypertension (RECOMPENSE)
Acronym: RECOMPENSE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Harm Jan Bogaard, Professor of Experimental Pulmonary Medicine, VU University of Amsterdam
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-512543-23-00; 2024-512543-23-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Arterial Hypertension PAH; Pulmonary Arterial Hypertension WHO Group I; Pulmonary Arterial Hypertension
Keywords: Pulmonary arterial hypertension; PAH; Right Ventricle; Sotatercept
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — ACE-011

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sotatercept treatment (Experimental): PAH patients receiving subcutaneous sotatercept injection
  Interventions: Drug: Sotatercept

INTERVENTIONS:
Drug: Sotatercept — Participants will receive open label subcutaneous sotatercept (starting dose, 0.3 mg per kilogram of body weight; target dose, 0.7 mg per kilogram) for 24 weeks

SUMMARY:
Pulmonary arterial hypertension (PAH) is a progressive disease characterized by vascular remodelling resulting in elevated pressures in the pulmonary artery (PA). This elevated pressure ultimately leads to fulminant right heart failure. Current therapeutic options are limited and are centred around vasodilatory medications such as phosphodiesterase-5 inhibitors and prostacyclin. While these medications allow for the widening of blood vessels that are narrowed due to remodelling, they have no effect on the remodelling itself.

Sotatercept is a novel medication which targets the BMPR2/TGF-β pathway and restore a pro- and anti- proliferative balance to ultimately counteract vascular remodelling. Recent phase 2 and 3 trials showed that treatment with sotatercept led to lower resistance and pressure in the pulmonary vasculature and improved exercise tolerance. However, these results were not coupled with an increase in cardiac output, a change that is seen with other PAH-medications with a primarily vasodilatory effect. These results suggest that cardiac work is reduced and cardiac efficiency is improved in patients being treated with sotatercept, in contrast with conventional PAH therapies. This is a potentially beneficial effect that may result in improved disease control in the long-term. Our study aims to explore the effect of sotatercept on cardiac work and function. We hypothesize that the effects of sotatercept are more beneficial for cardiac function than that of traditional PAH medications.

All participants included in the trial will undergo a screening visit in which it will be checked that all inclusion criteria and no exclusion criteria are met. The screening visit involves a physical exam, blood draw, 6-minute walk test, right heart catheterization (RHC) and cardiac magnetic resonance imaging (cMRI) with contrast to assess fibrosis.

Upon inclusion, all participants will receive a subcutaneous injection of sotatercept starting at a dose of 0.3 mg/kg. Participants will return to the hospital every three weeks for a blood draw, physical examination and an adverse event review. If the laboratory values (specifically haemoglobin and platelet counts) stay stable after the first dose, the dosage will be escalated to 0.7 mg/kg. The dose will not be escalated beyond 0.7 mg/kg.

After 24 weeks of receiving sotatercept, there will be an end of treatment visit including a physical exam, 6-minute walk test, right heart catheterization (RHC) and cardiac magnetic resonance imaging (cMRI) with contrast material.

DETAILED DESCRIPTION:
Recent phase 2 and phase 3 studies showed that treatment of PAH patients with the Activin ligand trap sotatercept results in significant reductions in PVR in addition to improvements in exercise capacity, as measured by 6MWD, and other clinical outcomes while effects on cardiac output were only minimal.

Assessment of intrinsic RV function is essential to understanding the effects of sotatercept on the myocardium. In order to make this assessment in a load-independent fashion, pressure-volume loops must be used. RV-PA coupling, the relationship between RV end systolic elastance and pulmonary arterial elastance, describes the relationship between RV contractility and RV afterload. The preservation of RV function rests on the delicate balance of RV coupling. In order to preserve RV function in PAH, an increase in afterload will be met with increased RV contractility. Uncoupling occurs in PAH when RV contractility fails to increase to match an elevated afterload leading to maladaptation and RV failure. Decreases in mPAP typically lead to decreases in RV contractility while exercise or sympathetic stimulation will lead to increased contractility.

This is a prospective, single center, single-arm, open-label, phase 4 study to evaluate the effects of sotatercept on RV function and dimensions in PAH. Twenty PAH patients will be enrolled at the Amsterdam UMC and receive open label subcutaneous sotatercept (starting dose, 0.3 mg per kilogram of body weight; target dose, 0.7 mg per kilogram) for 24 weeks. After signing informed consent and completion of screening, and before receiving the first drug dose, patients undergo right heart catheterization (RHC), and cMRI to determine pump function graphs and cardiac volumes and RV fibrosis. These procedures are repeated after the end of the treatment (EOT). The treatment period starts with the first dose of IMP and ends on the last day of IMP which is the day of the last dose of IMP at premature discontinuation or at week 24 ± 7 days. There is an additional follow-up period of 5 weeks after study completion.

Patients enrolled in the study will receive subcutaneous sotatercept (starting dose, 0.3 mg per kilogram of body weight; target dose, 0.7 mg per kilogram) for 24 weeks. After giving informed consent and before receiving the first drug dose, patients undergo RHC and cMRI to determine pump function graphs and cardiac volumes and assess fibrosis. Additionally, patients will undergo a physician assessment and blood sampling. All of these procedures will be repeated at the end of the treatment (EOT) visit after 24 weeks.

Recent phase 2 and phase 3 studies showed that treatment of pulmonary arterial hypertension (PAH) patients with the activin ligand trap sotatercept results in significant reductions in pulmonary vascular resistance (PVR) in addition to improvements in exercise capacity, as measured by the six minute walk distance (6MWD), and other clinical outcomes while effects on cardiac output (CO) are only minimal. These results contrast sharply with the results of studies with other PAH specific drugs, in which improvements in 6MWD were always reflected by profound increases in cardiac output. The fact that resting cardiac output after sotatercept treatment is not increased, may partly be attributed to a concomitant increase in blood hemoglobin levels, allowing a lower cardiac output to preserve oxygen delivery to the tissues. Moreover, conventional PAH drugs are not entirely pulmonary specific and cause systemic vasodilation, requiring an increase in cardiac output to maintain systemic blood pressure. In contrast, a slight increase in systemic blood pressure was observed in PAH patients treated with sotatercept. Considering these fundamental differences resulting from treatment with sotatercept, we hypothesize that the effects of sotatercept on cardiac function are much more beneficial than the effects of conventional PAH specific drugs.

This is a prospective, single center, single-arm, open-label, phase 4 study to evaluate the effects of sotatercept on RV function and dimensions in PAH. Twenty PAH patients will be enrolled at the Amsterdam UMC and receive open label subcutaneous sotatercept (starting dose, 0.3 mg per kilogram of body weight; target dose, 0.7 mg per kilogram) for 24 weeks

Patients enrolled in the study will receive subcutaneous sotatercept (starting dose, 0.3 mg per kilogram of body weight; target dose, 0.7 mg per kilogram) for 24 weeks. After giving informed consent and before receiving the first drug dose, patients undergo RHC and cMRI to determine pump function graphs and cardiac volumes and assess fibrosis. Additionally, patients will undergo a physician assessment and blood sampling. All of these procedures will be repeated at the end of the treatment (EOT) visit after 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients between 18-70 years of age
2. Able to provide signed informed consent
3. WHO FC II to IV
4. NTproBNP > 300 ng/L
5. PAH etiology belonging to one of the following groups (Nice classification):

   * Idiopathic PAH
   * Heritable PAH
6. Hemodynamic diagnosis of PAH confirmed by RHC during screening showing:

   * mPAP > 20 mmHg
   * Pulmonary capillary wedge pressure (PCWP) or left ventricular end diastolic pressure (LVEDP) ≤ 15 mmHg
   * PVR ≥ 4WU (320 dyn.sec.cm-5)
7. For patients treated with oral diuretics, treatment dose must have been stable at least 1 month prior to RHC during the screening period
8. All patients are on stable background therapy at least 3 months prior to RHC during the screening period
9. Women of childbearing potential must have a negative pregnancy test at screening and agree to use reliable methods of contraception
10. Males must agree to use a condom during sexual contact with a pregnant female or female of childbearing potential while participating in the study. Males should refrain from donating blood or sperm for the duration for the study and for 16 weeks after last dose of sotatercept

Exclusion Criteria:

1. Any contraindication to treatment with sotatercept
2. Body weight < 40 kg
3. Body mass index (BMI) > 35kg/m2
4. Pregnancy, breastfeeding, or intention to become pregnant during the study
5. Recently started (< 8 weeks prior to informed consent signature) or planned cardio-pulmonary rehabilitation program
6. Known concomitant life-threatening disease with a life expectancy < 12 months
7. Any condition likely to affect protocol or treatment compliance
8. Hospitalization for PAH within 3 months prior to informed consent signature
9. Left atrial volume per body surface area ≥ 43mL/m2 by echocardiography or CMR
10. Valvular disease grade 2 or higher
11. History of pulmonary embolism or deep vein thrombosis
12. Documented moderate to severe chronic obstructive pulmonary disease
13. Documented moderate to severe restrictive lung disease
14. Historical evidence of significant coronary artery disease
15. Diabetes mellitus
16. Active cancer
17. Systolic blood pressure < 90 mmHg
18. Need for dialysis
19. Responders to acute vasoreactivity testing based on medical history
20. Treatment with another investigational drug (planned, or taken within the 3 months prior to study treatment initiation)
21. Claustrophobia
22. Permanent cardiac pacemaker, automatic internal cardioverter
23. Metallic implant (e.g. defibrillator, neurostimulator, hearing aid, infusion device)
24. Atrial fibrillation, multiple premature ventricular or atrial contractions , or any other condition that would interfere with proper cardiac gating during CMR.
25. History of major bleeding
26. Hemoglobin above ULN for age and gender

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Power per beat | From enrollment to end of study at 24 weeks
  mean pulmonary arery pressure (mPAP) x stroke volume (SV)
Right ventricular pulmonary artery coupling | From enrollment to end of study at 24 weeks
  End systolic elastance (Ees)/ Arterial elastance (Ea) as derived from pressure-volume loops using right heart catheterization

SECONDARY OUTCOMES:
Right ventricular end systolic volume | From enrollment to the end of study at 24 weeks
  Right ventricular end systolic volume as measured by cardiac magnetic resonance imaging
Right ventricular end diastolic volume | From enrollment to the end of study at 24 weeks
  Right ventricular end diastolic volume as measured by cardiac magnetic resonance imaging
Right ventricular ejection fraction | From enrollment to the end of study at 24 weeks
  Right ventricular ejection fraction as measured by cardiac magnetic resonance imaging
Right ventricular mass | From enrollment to the end of study at 24 weeks
  Right ventricular mass as measured by cardiac magnetic resonance imaging
Stroke volume | From enrollment to the end of study at 24 weeks
  Stroke volume as measured by cardiac magnetic resonance imaging derived aortic flow
Left ventricular end diastolic volume | From enrollment to the end of study at 24 weeks
  Left ventricular end diastolic volume as measured by cardiac magnetic resonance imaging
Left ventricular end systolic volume | From enrollment to the end of study at 24 weeks
  Left ventricular end systolic volume as measured by cardiac magnetic resonance imaging
Left ventricular ejection fraction | From enrollment to the end of study at 24 weeks
  Left ventricular ejection fraction as measured by cardiac magnetic resonance imaging
Left ventricular mass | From enrollment to the end of study at 24 weeks
  Left ventricular mass as measured by cardiac magnetic resonance imaging
End-systolic elastance (Ees) | From enrollment to the end of study at 24 weeks
  End systolic elastance measured using pressure-volume loops derived from right heart catheteriazation
Arterial elastance (Ea) | From enrollment to the end of study at 24 weeks
  Arterial elastance measured using pressure-volume loops derived from right heart catheteriazation
End-diastolic elastance (Eed) | From enrollment to the end of study at 24 weeks
  End-diastolic elastance measured using pressure-volume loops derived from right heart catheteriazation
Right ventricular fibrosis | From enrollment to the end of study at 24 weeks
  Righ ventricular fibrosis derived from extracellular volume measurements using Modified Look-Locker inversion recovery MRI sequence

CONTACTS AND LOCATIONS:
Overall Officials: Harm Jan Bogaard, M.D., PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, location VUMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
A decision regarding data sharing will be made upon opening the study due to privacy concerns

REFERENCES:
- [Background] Vonk Noordegraaf A, Westerhof BE, Westerhof N. The Relationship Between the Right Ventricle and its Load in Pulmonary Hypertension. J Am Coll Cardiol. 2017 Jan 17;69(2):236-243. doi: 10.1016/j.jacc.2016.10.047. PMID 28081831
- [Background] Sniderman AD, Fitchett DH. Vasodilators and pulmonary arterial hypertension: the paradox of therapeutic success and clinical failure. Int J Cardiol. 1988 Aug;20(2):173-81. doi: 10.1016/0167-5273(88)90261-6. No abstract available. PMID 3061937
- [Background] Joshi SR, Liu J, Bloom T, Karaca Atabay E, Kuo TH, Lee M, Belcheva E, Spaits M, Grenha R, Maguire MC, Frost JL, Wang K, Briscoe SD, Alexander MJ, Herrin BR, Castonguay R, Pearsall RS, Andre P, Yu PB, Kumar R, Li G. Sotatercept analog suppresses inflammation to reverse experimental pulmonary arterial hypertension. Sci Rep. 2022 May 12;12(1):7803. doi: 10.1038/s41598-022-11435-x. PMID 35551212
- [Background] Gomberg-Maitland M, McLaughlin VV, Badesch DB, Ghofrani HA, Hoeper MM, Humbert M, Preston IR, Souza R, Waxman AB, de Oliveira Pena J, Lu JT, Manimaran S, Gibbs JSR. Long-Term Effects of Sotatercept on Right Ventricular Function: Results From the PULSAR Study. JACC Heart Fail. 2023 Oct;11(10):1457-1459. doi: 10.1016/j.jchf.2023.05.030. Epub 2023 Jul 12. No abstract available. PMID 37452806
- [Background] Souza R, Badesch DB, Ghofrani HA, Gibbs JSR, Gomberg-Maitland M, McLaughlin VV, Preston IR, Waxman AB, Grunig E, Kopec G, Meyer G, Olsson KM, Rosenkranz S, Lin J, Johnson-Levonas AO, de Oliveira Pena J, Humbert M, Hoeper MM. Effects of sotatercept on haemodynamics and right heart function: analysis of the STELLAR trial. Eur Respir J. 2023 Sep 21;62(3):2301107. doi: 10.1183/13993003.01107-2023. Print 2023 Sep. PMID 37696565
- [Background] Hoeper MM, Badesch DB, Ghofrani HA, Gibbs JSR, Gomberg-Maitland M, McLaughlin VV, Preston IR, Souza R, Waxman AB, Grunig E, Kopec G, Meyer G, Olsson KM, Rosenkranz S, Xu Y, Miller B, Fowler M, Butler J, Koglin J, de Oliveira Pena J, Humbert M; STELLAR Trial Investigators. Phase 3 Trial of Sotatercept for Treatment of Pulmonary Arterial Hypertension. N Engl J Med. 2023 Apr 20;388(16):1478-1490. doi: 10.1056/NEJMoa2213558. Epub 2023 Mar 6. PMID 36877098
- [Background] Humbert M, McLaughlin V, Gibbs JSR, Gomberg-Maitland M, Hoeper MM, Preston IR, Souza R, Waxman AB, Ghofrani HA, Escribano Subias P, Feldman J, Meyer G, Montani D, Olsson KM, Manimaran S, de Oliveira Pena J, Badesch DB. Sotatercept for the treatment of pulmonary arterial hypertension: PULSAR open-label extension. Eur Respir J. 2023 Jan 6;61(1):2201347. doi: 10.1183/13993003.01347-2022. Print 2023 Jan. PMID 36041750
- [Background] Humbert M, McLaughlin V, Gibbs JSR, Gomberg-Maitland M, Hoeper MM, Preston IR, Souza R, Waxman A, Escribano Subias P, Feldman J, Meyer G, Montani D, Olsson KM, Manimaran S, Barnes J, Linde PG, de Oliveira Pena J, Badesch DB; PULSAR Trial Investigators. Sotatercept for the Treatment of Pulmonary Arterial Hypertension. N Engl J Med. 2021 Apr 1;384(13):1204-1215. doi: 10.1056/NEJMoa2024277. PMID 33789009
- [Background] Handoko ML, de Man FS, Allaart CP, Paulus WJ, Westerhof N, Vonk-Noordegraaf A. Perspectives on novel therapeutic strategies for right heart failure in pulmonary arterial hypertension: lessons from the left heart. Eur Respir Rev. 2010 Mar;19(115):72-82. doi: 10.1183/09059180.00007109. PMID 20956170
- [Background] Messroghli DR, Radjenovic A, Kozerke S, Higgins DM, Sivananthan MU, Ridgway JP. Modified Look-Locker inversion recovery (MOLLI) for high-resolution T1 mapping of the heart. Magn Reson Med. 2004 Jul;52(1):141-6. doi: 10.1002/mrm.20110. PMID 15236377
- [Background] Waxman AB, Systrom DM, Manimaran S, de Oliveira Pena J, Lu J, Rischard FP. SPECTRA Phase 2b Study: Impact of Sotatercept on Exercise Tolerance and Right Ventricular Function in Pulmonary Arterial Hypertension. Circ Heart Fail. 2024 May;17(5):e011227. doi: 10.1161/CIRCHEARTFAILURE.123.011227. Epub 2024 Apr 4. PMID 38572639